CLINICAL TRIAL: NCT06682052
Title: Stress Ball Application on Pap Smear Test
Brief Title: Stress Ball Application on Anxiety and Pain During Pap Smear Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Dr., Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pap_smear_test; Hitit Uni Non-Interventional (Registry Identifier: Ethics Committee)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pain Management
Keywords: pap smear; anti stress ball; pain; anxiety
MeSH Terms: conditions — Agnosia; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): After obtaining the consent of the women, the Personal Information Form and the State Anxiety Inventory (STAI) will be filled out and prepared for the examination. The examination table is a stirrup table suitable for examination in the lithotomy position. It can be adjusted according to the height of the woman. When the women are taken to the examination table, a cover will be placed to protect privacy. No intervention other than routine application will be made to the women in the control group. After the Pap smear test is completed, the "State Anxiety Inventory (STAI)" and the "Visual Analog Scale (VAS)" will be applied.
- Group to be applied anti-stress ball (Experimental): After the women's consent is obtained, the Personal Information Form and State Anxiety Inventory (STAI) will be filled out and prepared for the examination. The examination table is a stirrup table suitable for examination in the lithotomy position. It can be adjusted according to the woman's height. When the women are taken to the examination table, a cover will be placed to protect privacy.
  The women will be given a round, silicone, medium-sized and medium-hard anti-stress ball, and they will be told how to use the stress ball, and they will be asked to squeeze the anti-stress ball throughout the examination, allowing the patients to rest occasionally as they wish. The women will be told to count to 3 as they squeeze the anti-stress ball, then to relax the stress ball and repeat this process.
  After the Pap smear test is completed, the "State Anxiety Inventory (STAI)" and the "Visual Analog Scale (VAS)" will be applied.
  Interventions: Other: anti-stress ball

INTERVENTIONS:
Other: anti-stress ball — The women will be given a round, silicone, medium-sized and medium-hard anti-stress ball, and they will be told how to use the stress ball, and they will be asked to squeeze the anti-stress ball throughout the examination, allowing the patients to rest occasionally as they wish. The women will be told to count to 3 as they squeeze the anti-stress ball, then to relax the stress ball and repeat this process.
  Arms: Group to be applied anti-stress ball

SUMMARY:
A negative pelvic examination experience may deter women from returning for follow-up tests, thus reducing the intended benefit of gynecological screening. For all these reasons, women's experiences with pelvic examinations and related conditions should be taken into account by healthcare services. Although the pelvic examination is relatively brief, cognitive-behavioral interventions that focus or distract the patient's attention have been shown to be effective in reducing pain and anxiety during brief medical interventions. Reducing pain and anxiety during medical procedures is an important factor in patient satisfaction. Although there are many methods to reduce stress, it is thought that the inexpensive and easily accessible anti-stress ball can be used as a distraction method. A study has determined that a stress ball reduces anxiety and pain during angiography. No studies were found in the literature examining the effects of an anti-stress ball on anxiety and pain during a pelvic examination.

DETAILED DESCRIPTION:
Pelvic examination is a common approach to evaluate a woman's external and internal genitalia and pelvic organs. Pelvic examination is usually performed during gynecological health checks; as part of the diagnosis, treatment, and follow-up of gynecological problems (e.g., sexually transmitted infections, genital cancer, pap smear test); and during perinatal care. Although women usually have a pelvic examination at least once in their lifetime, they avoid having further pelvic examinations due to fear that their privacy may be compromised. Women often experience fear, anxiety, and pain during pelvic examinations. Studies also show that women experience pelvic examinations as uncomfortable, intrusive, embarrassing, humiliating, and upsetting. A study conducted in Turkey reported that women experienced intense anxiety during a pelvic examination and that the most important reason for anxiety was the disruption of privacy. A study conducted in Denmark reported that 75% of women experienced negative emotions during a pelvic examination. Similarly, a study conducted in the Netherlands reported that women felt pain and embarrassment during a pelvic examination, were unable to relax, and were treated disrespectfully. Women may be embarrassed by the exposure of their genitals, a bad smell, or looking dirty during the examination. On the other hand, they may fear that a pathological condition may be discovered. Losing control over their bodies and giving information about their sexual habits are also noteworthy among other reasons for anxiety. Patient-related risk factors for a negative pelvic examination experience include young age, having a male examiner, receiving negative information from peers, previous negative experiences during a pelvic examination, religious and cultural beliefs, and most importantly, a history of sexual trauma. Healthcare provider-related factors that contribute to a negative pelvic examination experience include performing the pelvic examination hastily, insensitively, and without proper explanations. A trusting relationship between the healthcare provider and patients is a mitigating factor to reduce the negative pelvic examination experience. A negative pelvic examination experience may deter women from returning for follow-up tests, thereby reducing the intended benefit of gynecologic screening. For all these reasons, women's experiences with pelvic examinations and related conditions should be taken into account by healthcare services. Although the pelvic examination is relatively brief, cognitive-behavioral interventions that focus or distract the patient's attention have been shown to be effective in reducing pain and anxiety during brief medical interventions. Reducing pain and anxiety during medical procedures is an important factor in patient satisfaction. Although there are many methods of reducing stress, it is thought that the inexpensive and easily accessible anti-stress ball can be used as a method of distraction. In one study, it was determined that the stress ball reduced anxiety and pain during angiography.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over,
* At least primary school graduates,
* Not pregnant,
* Married,
* No physical obstacles to using the anti-stress ball,
* Those who agree to participate in the study.

Exclusion Criteria:

* Acute pelvic pain,
* Any injury or lesion to the perineum that may cause pain during the examination,
* Analgesic or anxiolytic use within 24 hours before the examination,
* Vaginismus,
* History of sexual abuse,
* History of a traumatic pelvic examination.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | during application (average 2nd minute)
  Visual Analog Scale for pain

SECONDARY OUTCOMES:
State Anxiety Inventory (STAI): | after and before procedure (average 5nd minute before and after)
  It was designed by Spielberger et al. (1983) to measure state anxiety, which refers to how one feels at the moment, and trait anxiety, which refers to how one feels in general. The State Anxiety Inventory consists of 20 self-reported 4-point Likert-type items, with negatively worded items reverse scored. Total scores range from 20 to 80, with higher scores indicating increased levels of anxiety. The Turkish adaptation of the scale was made by Öner and Le Compte (1983). In studies conducted with different samples, reliability coefficients of the State Anxiety Inventory have been reported between 0.83 and 0.92.

IPD SHARING:
Plan to Share IPD: No